CLINICAL TRIAL: NCT00221234
Title: The Development and Evaluation of Physical Activity Behavioural Strategies for Adults With Type 2 Diabetes: A Population Based Approach
Brief Title: Alberta Diabetes and Physical Activity Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MOP-69070
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity

INTERVENTIONS:
Behavioral: Print materials, pedometers/logbooks
Behavioral: Print materials, pedometers/logbooks, telephone counselling

SUMMARY:
This project will assess the incremental and cumulative impact of three behavioural intervention strategies for the promotion of physical activity in the adult general population with Type 2 diabetes.

DETAILED DESCRIPTION:
An increasing prevalence of Type 2 Diabetes is associated with the aging population, a significant rise in the prevalence of obesity, and a sedentary lifestyle. In Canada, 4.9-7.0% over the age of 12 and 17% over the age of 64 are estimated to have diabetes, 90-95% of which will be Type 2. Strong evidence supports the importance of physical activity in the management of Type 2 Diabetes. However, current literature lacks clear understanding of best strategies for physical activity behaviour change in this target population. Existing studies employ resource intensive, one-to-one individual and clinically-based approaches with limited theoretical grounding for recommended health behaviour change. Most fail to offer practical, sustainable, economically viable solutions, with documented long-term intervention efficacy. The call to move beyond the clinical focus by including theoretically population-based and "real-life" approaches for the management Type 2 Diabetes remains largely unheeded. The three interventions are: (1) standard print-based physical activity educational materials provided by the Canadian Diabetes Association (CDA); (2) CDA materials + pedometers and a log book + theoretical stage-matched print-based physical activity materials; and, (3) the same as intervention 2 with the addition of a 12-month physical activity telephone counseling protocol.

ELIGIBILITY:
Inclusion Criteria:

>18 years old, Type 2 Diabetes, Living in the province of Alberta, Can communicate in English.

Exclusion Criteria:

Serious Contraindications to Physical Activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Physical Activity Behaviour

SECONDARY OUTCOMES:
HbA1c, CRP, lipid concentrations, fasting blood glucose, insulin, health related quality of life, psychosocial predictors of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ron C Plotnikoff, PhD, Principal Investigator — University of Alberta

REFERENCES:
- [Derived] Plotnikoff RC, Karunamuni N, Courneya KS, Sigal RJ, Johnson JA, Johnson ST. The Alberta Diabetes and Physical Activity Trial (ADAPT): a randomized trial evaluating theory-based interventions to increase physical activity in adults with type 2 diabetes. Ann Behav Med. 2013 Feb;45(1):45-56. doi: 10.1007/s12160-012-9405-2. PMID 22922954
- [Derived] Plotnikoff RC, Courneya KS, Sigal RJ, Johnson JA, Birkett N, Lau D, Raine K, Johnson ST, Karunamuni N. Alberta Diabetes and Physical Activity Trial (ADAPT): a randomized theory-based efficacy trial for adults with type 2 diabetes--rationale, design, recruitment, evaluation, and dissemination. Trials. 2010 Jan 12;11:4. doi: 10.1186/1745-6215-11-4. PMID 20067626